CLINICAL TRIAL: NCT06507540
Title: Dental Emergencies Among Patients of the Health Care Access Center at the University Hospital of Nancy
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Baudet Alexandre, Dental hospital practitioner and associate professor (MCU-PH), Central Hospital, Nancy, France
Other Study IDs: 2024PI135
Record Dates: First submitted 2024-07-06; First posted 2024-07-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Community Dentistry; Emergencies
Keywords: Dentistry; Dental care
MeSH Terms: conditions — Emergencies | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (observational study) — Retrospective description of diagnostics and treatements of dental emergencies

SUMMARY:
The dental Health Care Access Center at the University Hospital of Nancy opened in January 2023. The patients ot the dental Health Care Access Center consulting the dental department have largely been treated as dental emergencies. However, to date, no study has been carried out into the nature of these patients' consultations or treatments. This new patient management has necessitated adaptations within the dental department, but there are no data to enable us to better understand and organize the care of these patients. Moreover, the cost of dental emergencies has not been estimated.

Our hypotheses are that patients of the dental Health Care Access Center consulted mainly the dental departement for painful emergencies and that the emergency dental cares were provided rapidly and at low cost. On the other hand, patient flow was probably correlated with the days when a social worker of the dental Health Care Access Center was present, referring patients to the dental department.

The main aim of the study is to describe the nature of emergency dental care provided to patients of the dental Health Care Access Center at the dental department of the University Hospital of Nancy.

The secondary objectives are: i) to describe the temporality of dental emergency consultations for patients of the dental Health Care Access Center, ii) to describe the rate of dental consultations secondary to an initial emergency consultation, and iii) describe the direct cost of emergency consultations and treatment.

DETAILED DESCRIPTION:
In France, the Health Care Access Center are gateway medical and social services for people who need healthcare but have difficulty accessing it due to lack of social protection, living conditions or financial difficulties. They provide access to medical and dental consultations. The development of dental Health Care Access Center across France is helping to improve the territorial coverage of primary care services. Consultations, diagnostic and treatments are provided free of charge to patients of the Health Care Access Center.

ELIGIBILITY:
Inclusion Criteria:

* All patients from the dental Health Care Access Center who consulted for a dental emergency at the dental department of the University Hospital of Nancy from 1st January 2023 to 30 June 2024.

Exclusion Criteria:

* Patient who has objected to the use of his or her medical data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients from the dental Health Care Access Center who consulted for a dental emergency at the dental department of the University Hospital of Nancy
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dental care reported in the medical record | 18 months
  Types of emergency dental care parformed among patients referred by the Health Care Access Center at the dental service of the University Hospital of Nancy

SECONDARY OUTCOMES:
Days of dental emergencies | 18 months
  Month and day of the week of emergency consultations for patients of the dental Health Care Access Center
Follow-up | 18 months
  Number and delay of dental consultations in the dental service following an initial emergency consultation
Costs | 18 months
  Cost of consultations and treatments performed at the dental service

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France